CLINICAL TRIAL: NCT03805217
Title: Prospective, Single-Arm, Open-Label, Multicenter Study of Hypotension Prevention and Treatment in Patients Receiving Arterial Pressure Monitoring with Acumen™ Hypotension Prediction Index Feature Software
Brief Title: Hypotension Prediction Index Study (HPI Study)
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-15
Record Dates: First submitted 2019-01-14; First posted 2019-01-15 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2020-08

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: EV1000A Clinical Platform with Acumen Hypotension Prediction Index Feature Software — EV1000A Clinical Platform with Acumen Hypotension Prediction Index Feature Software

SUMMARY:
A prospective, single-arm, open-label, multicenter post-approval study to determine whether the use of the Acumen HPI Software to guide intraoperative hemodynamic management in non-cardiac surgery reduces the duration of intraoperative hypotension below a threshold of Mean Arterial Pressure (MAP)

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent;
2. Age ≥ 18 years;
3. ASA Physical Status 3 or 4;
4. Moderate- or high-risk non-cardiac surgery (for example, orthopedic, spine, urology, and general surgery);
5. Planned pressure monitoring with an arterial line;
6. General anesthesia;
7. Surgery duration expected to last ≥ 3 hours from induction;
8. Planned overnight hospitalization.

Exclusion Criteria:

1. Participating in another (interventional) study;
2. Contraindication to the invasive blood pressure monitoring;
3. Patient who is confirmed to be pregnant and/or nursing mothers;
4. Emergency surgery;
5. Known clinically important intra-cardiac shunts;
6. Patient in whom an intraoperative MAP target will be < 65 mmHg;
7. Known aortic stenosis with valve area ≤ 1.5 cm2;
8. Known moderate to severe aortic regurgitation;
9. Known moderate to severe mitral regurgitation;
10. Known moderate to severe mitral stenosis;
11. Patient or surgical procedure type known as an SVV limitation (5) (e.g. tidal volume <8mL/kg of theoretical ideal weight, spontaneous ventilation, persistent cardiac arrhythmia, known atrial fibrillation, open chest surgery, Heart Rate/Respiratory Rate (HR/RR) ratio <3.6);
12. Current persistent atrial fibrillation;
13. Known acute congestive heart failure;
14. Craniotomy;
15. Surgery duration expected to last < 3 hours;
16. Burn surgeries;
17. Patients with an intra-aortic balloon pump (IABP) or ventricular assist device(s);
18. Patient transfer from ICU requiring multiple vasoactive agents and known diagnosis of ongoing active sepsis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects recruited and enrolled should be classified as American Society of Anesthesiologist (ASA) physical status 3-4 who are scheduled for moderate-to-high-risk non-cardiac surgery and will be receiving pressure monitoring with an arterial line. Potentially qualifying patients will be evaluated during their preoperative anesthesia clinic visits.
Sampling Method: Probability Sample
Enrollment: 485 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Reduction of Intraoperative Hypotension | Duration of Surgery
  Duration (t [min]) reduction of intraoperative hypotension (defined as MAP < 65 mmHg for at least 1 minute) as compared with a historic retrospective control group

SECONDARY OUTCOMES:
Intraoperative Hypotension in Each Subject | Duration of Surgery
  The determination of total area under the curve (time and MAP) for Intraoperative Hypotension in each subject. This endpoint is correlated with the duration and a descriptive analysis of this endpoint will be presented with the mean, standard deviation, median, minimum and maximum.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Abdelnour, MS, BSN, Study Director — Edwards Lifesciences
Locations (11):
- United States (11):
  - Stanford Health Care, Stanford, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bao X, Kumar SS, Shah NJ, Penning D, Weinstein M, Malhotra G, Rose S, Drover D, Pennington MW, Domino K, Meng L, Treggiari M, Clavijo C, Wagener G, Chitilian H, Maheshwari K; HPI Study Team. AcumenTM hypotension prediction index guidance for prevention and treatment of hypotension in noncardiac surgery: a prospective, single-arm, multicenter trial. Perioper Med (Lond). 2024 Mar 4;13(1):13. doi: 10.1186/s13741-024-00369-9. PMID 38439069